CLINICAL TRIAL: NCT02021188
Title: The Vascular Inflammation Imaging Using Somatostatin Receptor Positron Emission Tomography Study
Brief Title: Vascular Inflammation Imaging Using Somatostatin Receptor Positron Emission Tomography
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, James Rudd, HEFCE Senior Lecturer and Honorary Consultant Cardiologist, University of Cambridge
Other Study IDs: A093095
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Atherosclerosis; Stroke; Transient Ischemic Attack; Chronic Stable Angina; Acute Coronary Syndrome
Keywords: Vascular inflammation; Atherosclerosis; Positron Emission Tomography; Molecular Imaging; 68Ga-DOTATATE
MeSH Terms: conditions — Atherosclerosis; Stroke; Ischemic Attack, Transient; Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Carotid artery plaques
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carotid artery disease: Participants with symptomatic or asymptomatic carotid artery plaques
- Coronary artery disease: Participants with stable coronary artery disease or recent acute coronary syndrome

SUMMARY:
This VISION study aims to investigate the role of inflammation in atherosclerosis using 68Ga- DOTATATE PET, and to validate 68Ga-DOTATATE PET imaging for the detection and quantification of vascular inflammation in the aorta, coronary and carotid arteries. This study will test the hypothesis that in subjects undergoing carotid endarterectomy for symptomatic plaques, there will be a positive correlation between carotid artery 68Ga-DOTATATE PET signal and the underlying degree of carotid inflammation measured by immunohistochemical analysis.

DETAILED DESCRIPTION:
Clinical events in atherosclerosis are largely driven by inflammation. Molecular imaging of atherosclerosis can potentially identify high-risk lesions, help guide treatment and illuminate the underlying biology of the disease. 18F-fluorodeoxyglucose (18F-FDG) PET is the gold-standard nuclear molecular imaging technique with well-established roles in atherosclerosis imaging. However, the arterial 18F-FDG signal is non-specific, although it is related to increased macrophage activity with contributions from hypoxia and angiogenesis. Coronary artery imaging with 18F-FDG is particularly difficult, mainly due to high background myocardial cell 18F-FDG uptake, which obscures interpretation of the coronary signal. Efforts to suppress myocardial 18F-FDG uptake with dietary manipulation are challenging for patients and have limited efficacy.

PET tracers currently used in cancer imaging, such as 68Ga-DOTATATE, are potentially more specific for inflammation and also lack myocardial muscle uptake. 68Ga-DOTATATE might therefore be better suited than 18F-FDG for imaging inflammation, particularly within the coronary arteries. The VISION study is a prospective, observational study designed to investigate the biology of plaque inflammation in atherosclerosis, using PET imaging with the somatostatin receptor ligand 68Ga-DOTATATE. 50 subjects with atherosclerosis will undergo sequential PET/CT imaging with 68Ga-DOTATATE and 18F-FDG, along with contrast angiography of the carotid and coronary arteries. Autoradiography and immunohistochemistry of excised carotid plaques will be used to validate the imaging data. If successful, 68Ga-DOTATATE imaging will offer a cheaper, more specific non-invasive measure of inflammation than 18F- FDG, particularly in the coronary arteries. This opens up the possibility of better risk stratification for patients with atherosclerosis and could provide a non-invasive platform to test the effects of novel anti-atherosclerosis drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years of age
* Can provide written, fully informed consent
* Have had a transient ischemic attack (TIA) or stroke within the preceding four weeks due to carotid artery atherosclerosis; or have ≥30% carotid artery or epicardial coronary artery stenosis

Exclusion Criteria:

* Renal impairment (eGFR<30mls/min)
* History of contrast nephropathy
* Atrial fibrillation
* Any condition, in the opinion of the investigator, which prevents the participant from lying flat during scanning
* Women of childbearing potential
* Inability to provide written informed consent
* Haemorrhagic stroke within 3 months of study entry
* Total occlusion of a culprit carotid artery
* Any medical condition, vital sign or laboratory value that, in the opinion of the investigator, makes the subject ineligible for inclusion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit participants with recent transient ischaemic attack or stroke due to carotid artery disease, from which they have made a good functional recovery. A proportion of these patients will undergo carotid endarterectmy as part of clinical management. We will also recruit participants with asymptomatic carotid atheroma, and those with stable coronary artery disease or recent acute coronary syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Correlation of 68Ga-DOTATATE PET signal to carotid plaque inflammation | Baseline
  This primary outcome measure is correlation between carotid artery 68Ga-DOTATATE PET signal (TBR) and the underlying degree of carotid inflammation, measured by CD68 immunohistochemistry, in patients undergoing carotid endarterectomy.

SECONDARY OUTCOMES:
Comparison of 68Ga-DOTATATE signal between symptomatic and asymptomatic carotid plaques | Baseline (<1 month from event)
Correlation of carotid artery and coronary artery 68Ga-DOTATATE uptake | Baseline
Correlation of Framingham Cardiovascular Risk Scores to arterial 68Ga-DOTATATE uptake | Baseline
Correlation between carotid artery 68Ga-DOTATATE autoradiographic signal and degree of carotid inflammation, measured by CD68 immunohistochemistry | Baseline
Comparison of myocardial 68Ga-DOTATATE and 18F-FDG uptake | Baseline (2 scans within 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: James HF Rudd, PhD, FRCP, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Tarkin JM, Calcagno C, Dweck MR, Evans NR, Chowdhury MM, Gopalan D, Newby DE, Fayad ZA, Bennett MR, Rudd JHF. 68Ga-DOTATATE PET Identifies Residual Myocardial Inflammation and Bone Marrow Activation After Myocardial Infarction. J Am Coll Cardiol. 2019 May 21;73(19):2489-2491. doi: 10.1016/j.jacc.2019.02.052. No abstract available. PMID 31097170
- [Derived] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306